CLINICAL TRIAL: NCT02275910
Title: A Phase 1 Study of E7090 in Subjects With Solid Tumor
Brief Title: Phase 1 Study of E7090 in Subjects With Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7090-J081-101
Record Dates: First submitted 2014-10-20; First posted 2014-10-27 (Estimated); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Tumors
Keywords: Solid Tumors; E7090
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- E7090 Arm (Experimental): Oral, starting dose 1 mg once a day, dose escalation in part 1. Cycle 0 is for 7 days. For Cycle 1 and onward, each cycle is 28 days long. The Cycle 0 is set up for PK analysis of a single dose of E7090. In the following Cycle 1, subjects will be administered E7090 QD, and the PK and safety will be assessed for 28 days. One or two doses may be selected from part 1 for Part 2. E7090 will be administered continuously once a daily. Subjects can continue treatment unless they meet discontinuation criteria.
  Interventions: Drug: E7090

INTERVENTIONS:
Drug: E7090

SUMMARY:
This is a Phase 1 study of E7090 in subjects with advanced solid tumors. This study will be conducted in 2 parts:

1. Part 1 will be the dose escalation portion of this study to determine the maximum tolerated dose in subjects with solid tumors, and
2. Part 2 will comprise cohort expansions to further characterize the safety and tolerability of E7090 and to assess preliminary efficacy of E7090 in subjects with solid tumors characterized by genetic abnormalities in FGF/FGFR pathway.

ELIGIBILITY:
Inclusion Criteria: Part 1and Part 2

1. Provide written informed consent
2. Male or female subjects age >= 20 years at the time of informed consent
3. Subjects with a histological and/or cytological diagnosis of solid tumor
4. Subjects who failed standard therapies, or for which no appropriate treatment is available.
5. Subjects with Performance Status (PS) score of 0-1 established by Eastern Cooperative Oncology Group (ECOG)
6. Subjects who are expected to survive for 3 months or longer after starting administration of the investigational drug.

   Inclusion Criteria: Part 2 only
7. Subjects with tumor expressing genetic abnormality in FGF/FGFR (fibroblast growth factor/ fibroblast growth factor receptor)pathway.

Exclusion criteria

1. Patients with brain metastasis who have clinical symptoms or requiring treatment.
2. Medical history of clinically significant cardiovascular impairment
3. Concomitant systemic infection requiring medical treatment
4. Effusion requiring drainage
5. Known intolerance to the study drug (or any of excipients)
6. Subjects whose toxicity of previous treatment has not recovered to Grade 1 or lower (except for alopecia).
7. Inability to take oral medication, or malabsorption syndrome, or any other uncontrolled gastrointestinal condition (e.g., nausea, diarrhea, or vomiting) that might impair the bioavailability of E7090.
8. Psychiatric disorder (e.g., alcohol or drug dependency) judged to be ineligible for study entry by the investigator or subinvestigator
9. Females who are pregnant or breastfeeding
10. Any subjects who are judged by the principal investigator or the other investigators to be inappropriate as subjects in this clinical study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10-28 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- Japan (18):
  - Eisai Trial Site #1, Nagoya, Aichi-ken
  - Eisai Trial Site #1, Kashiwa, Chiba
  - Eisai Trial Site #1, Matsuyama, Ehime
  - Eisai Trial Site #1, Sapporo, Hokkaido
  - Eisai Trial Site #1, Amagasaki, Hyōgo
  - Eisai Trial Site #1, Tsukuba, Ibaraki
  - Eisai Trial Site #1, Kawasaki, Kanagawa
  - Eisai Trial Site #1, Yokohama, Kanagawa
  - Eisai Trial Site #1, Chuo-ku, Niigata
  - Eisai Trial Site #1, Kitaadachi, Saitama
  - Eisai Trial Site #1, Chuo-Ku, Tokyo
  - Eisai Trial Site #1, Koto-ku, Tokyo
  - Eisai Trial Site #1, Chiba
  - Eisai Trial Site #1, Fukuoka
  - Eisai Trial Site #1, Kyoto
  - Eisai Trial Site #1, Osaka
  - Eisai Trial Site #2, Osaka
  - Eisai Trial Site #3, Osaka

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 18 investigative sites in Japan from 28 October 2014 to 03 September 2021.
Pre-assignment Details: A total of 40 participants were enrolled in this study. This study consisted of two parts: Part 1 and Part 2. In Part 1, 24 participants were enrolled and received study treatment and in Part 2, 16 participants were enrolled and received the study treatment.
Groups:
- Part 1: E7090 1 mg With Solid Tumor: Participants with solid tumor received E7090 1 milligram (mg) capsules orally, once on Day 1 of Cycle 0 (Cycle length=7 days) in the fasting state and thereafter once daily in Cycle 1 and 2 and subsequent cycles (Cycle length=28 days) unless withdrawal of consent, major inclusion/exclusion criteria violation, difficulty in continuing the study due to an adverse event, pregnancy, disease progression, dose reduction to <1 mg (Part 1) or <35 mg (Part 2) required due to an adverse drug reaction, other cases where the investigator or subinvestigator considers study discontinuation appropriate.
- Part 1: E7090 2 mg With Solid Tumor: Participants with solid tumor received E7090 2 mg capsules orally, once on Day 1 of Cycle 0 (Cycle length=7 days) in the fasting state and thereafter once daily in Cycle 1 and 2 and subsequent cycles (Cycle length=28 days) unless withdrawal of consent, major inclusion/exclusion criteria violation, difficulty in continuing the study due to an adverse event, pregnancy, disease progression, dose reduction to <1 mg (Part 1) or <35 mg (Part 2) required due to an adverse drug reaction, other cases where the investigator or subinvestigator considers study discontinuation appropriate.
- Part 1: E7090 4 mg With Solid Tumor: Participants with solid tumor received E7090 4 mg capsules orally, once on Day 1 of Cycle 0 (Cycle length=7 days) in the fasting state and thereafter once daily Cycle 1 and 2 and subsequent cycles (Cycle length=28 days) unless withdrawal of consent, major inclusion/exclusion criteria violation, difficulty in continuing the study due to an adverse event, pregnancy, disease progression, dose reduction to <1 mg (Part 1) or <35 mg (Part 2) required due to an adverse drug reaction, other cases where the investigator or subinvestigator considers study discontinuation appropriate.
- Part 1: E7090 8 mg With Solid Tumor: Participants with solid tumor received E7090 8 mg capsules orally, once on Day 1 of Cycle 0 (Cycle length=7 days) in the fasting state and thereafter once daily in 28-days treatment cycles for Cycle 1 and 2 and subsequent cycles unless withdrawal of consent, major inclusion/exclusion criteria violation, difficulty in continuing the study due to an adverse event, pregnancy, disease progression, dose reduction to <1 mg (Part 1) or <35 mg (Part 2) required due to an adverse drug reaction, other cases where the investigator or subinvestigator considers study discontinuation appropriate.
- Part 1: E7090 16 mg With Solid Tumor: Participants with solid tumor received E7090 16 mg capsules orally, once on Day 1 of Cycle 0 (Cycle length=7 days) in the fasting state and thereafter once daily in 28-days treatment cycles for Cycle 1 and 2 and subsequent cycles (Cycle length=28 days) unless withdrawal of consent, major inclusion/exclusion criteria violation, difficulty in continuing the study due to an adverse event, pregnancy, disease progression, dose reduction to <1 mg (Part 1) or <35 mg (Part 2) required due to an adverse drug reaction, other cases where the investigator or subinvestigator considers study discontinuation appropriate.
- Part 1: E7090 30 mg With Solid Tumor: Participants with solid tumor received E7090 30 mg capsules orally, once on Day 1 of Cycle 0 (Cycle length=7 days) in the fasting state and thereafter once daily in Cycle 1 and 2 and subsequent cycles (Cycle length=28 days) unless withdrawal of consent, major inclusion/exclusion criteria violation, difficulty in continuing the study due to an adverse event, pregnancy, disease progression, dose reduction to <1 mg (Part 1) or <35 mg (Part 2) required due to an adverse drug reaction, other cases where the investigator or subinvestigator considers study discontinuation appropriate.
- Part 1: E7090 60 mg With Solid Tumor: Participants with solid tumor received E7090 60 mg capsules orally, once on Day 1 of Cycle 0 (Cycle length=7 days) in the fasting state and thereafter once daily in Cycle 1 and 2 and subsequent cycles (Cycle length=28 days) unless withdrawal of consent, major inclusion/exclusion criteria violation, difficulty in continuing the study due to an adverse event, pregnancy, disease progression, dose reduction to <1 mg (Part 1) or <35 mg (Part 2) required due to an adverse drug reaction, other cases where the investigator or subinvestigator considers study discontinuation appropriate.
- Part 1: E7090 100 mg With Solid Tumor: Participants with solid tumor received E7090 100 mg capsules orally, once on Day 1 of Cycle 0 (Cycle length=7 days) in the fasting state and thereafter once daily in Cycle 1 and 2 and subsequent cycles (Cycle length=28 days) unless withdrawal of consent, major inclusion/exclusion criteria violation, difficulty in continuing the study due to an adverse event, pregnancy, disease progression, dose reduction to <1 mg (Part 1) or <35 mg (Part 2) required due to an adverse drug reaction, other cases where the investigator or subinvestigator considers study discontinuation appropriate.
- Part 1: E7090 140 mg With Solid Tumor: Participants with solid tumor received E7090 140 mg capsules orally, once on Day 1 of Cycle 0 (Cycle length=7 days) in the fasting state and thereafter once daily in Cycle 1 and 2 and subsequent cycles (Cycle length=28 days) unless withdrawal of consent, major inclusion/exclusion criteria violation, difficulty in continuing the study due to an adverse event, pregnancy, disease progression, dose reduction to <1 mg (Part 1) or <35 mg (Part 2) required due to an adverse drug reaction, other cases where the investigator or subinvestigator considers study discontinuation appropriate.
- Part 1: E7090 180 mg With Solid Tumor: Participants with solid tumor received E7090 180 mg capsules orally, once on Day 1 of Cycle 0 (Cycle length=7 days) in the fasting state and thereafter once daily in Cycle 1 and 2 and subsequent cycles (Cycle length=28 days) unless withdrawal of consent, major inclusion/exclusion criteria violation, difficulty in continuing the study due to an adverse event, pregnancy, disease progression, dose reduction to <1 mg (Part 1) or <35 mg (Part 2) required due to an adverse drug reaction, other cases where the investigator or subinvestigator considers study discontinuation appropriate.
- Part 2: E7090 140 mg With Gastric Cancer: Participants with gastric cancer received E7090 140 mg capsules orally, on Days 1 and 8 of Cycle 1 in the fasting state and subsequent cycles (Cycle length=28 days) unless withdrawal of consent, major inclusion/exclusion criteria violation, difficulty in continuing the study due to an adverse event, pregnancy, disease progression, dose reduction to <1 mg (Part 1) or <35 mg (Part 2) required due to an adverse drug reaction, other cases where the investigator or subinvestigator considers study discontinuation appropriate.
- Part 2: E7090 140 mg With Cholangiocarcinoma: Participants with Cholangiocarcinoma received E7090 140 mg capsules orally, on Days 1 and 8 of Cycle 1 in the fasting state and subsequent cycles (Cycle length=28 days) unless withdrawal of consent, major inclusion/exclusion criteria violation, difficulty in continuing the study due to an adverse event, pregnancy, disease progression, dose reduction to <1 mg (Part 1) or <35 mg (Part 2) required due to an adverse drug reaction, other cases where the investigator or subinvestigator considers study discontinuation appropriate.
Period: Overall Study
Arm/Group | Part 1: E7090 1 mg With Solid Tumor | Part 1: E7090 2 mg With Solid Tumor | Part 1: E7090 4 mg With Solid Tumor | Part 1: E7090 8 mg With Solid Tumor | Part 1: E7090 16 mg With Solid Tumor | Part 1: E7090 30 mg With Solid Tumor | Part 1: E7090 60 mg With Solid Tumor | Part 1: E7090 100 mg With Solid Tumor | Part 1: E7090 140 mg With Solid Tumor | Part 1: E7090 180 mg With Solid Tumor | Part 2: E7090 140 mg With Gastric Cancer | Part 2: E7090 140 mg With Cholangiocarcinoma
Started | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 3 | 10 | 6
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 10 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Not completed — Subject Choice | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Radiological Disease Progression | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set was the group of participants who received at least 1 dose of E7090.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: E7090 1 mg With Solid Tumor | Part 1: E7090 2 mg With Solid Tumor | Part 1: E7090 4 mg With Solid Tumor | Part 1: E7090 8 mg With Solid Tumor | Part 1: E7090 16 mg With Solid Tumor | Part 1: E7090 30 mg With Solid Tumor | Part 1: E7090 60 mg With Solid Tumor | Part 1: E7090 100 mg With Solid Tumor | Part 1: E7090 140 mg With Solid Tumor | Part 1: E7090 180 mg With Solid Tumor | Part 2: E7090 140 mg With Gastric Cancer | Part 2: E7090 140 mg With Cholangiocarcinoma | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 3 | 10 | 6 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (6.36) | 68.0 (5.66) | 57.5 (3.54) | 58.5 (23.33) | 58.5 (6.36) | 58.5 (6.36) | 71.0 (3.61) | 67.0 (1.00) | 64.0 (6.93) | 53.3 (11.93) | 67.5 (9.07) | 53.7 (10.65) | 62.5 (10.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 1 | 1 | 0 | 2 | 1 | 1 | 3 | 3 | 1 | 17
  Male | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 2 | 2 | 0 | 7 | 5 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 2 | 2 | 2 | 2 | 2 | 1 | 3 | 3 | 3 | 3 | 10 | 6 | 39
  Chinese | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 3 | 10 | 6 | 40

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: DLT was graded using Common Terminology Criteria for Adverse Events version 4.03 as follows: a. febrile neutropenia, or Grade 4 neutropenia persisting for greater than or equal to (>=) 7 days, b. Grade 4 thrombocytopenia, or Grade 3 thrombocytopenia requiring platelet transfusions, c. Grade >=3 non-hematological toxicity, except for: clinically insignificant laboratory abnormalities, toxicity Grade less than or equal to (<=) 2 by best supportive care; d. potentially clinically significant, new radiographic mineralization in soft tissue, kidneys, intestines, heart, lungs, or other organs; e. Hyperphosphatemia meeting either for: serum phosphate level greater than (>) 7 milligram per deciliter (mg/dL) persisting for >=7 days despite best treatment, serum phosphate level >9 mg/dL despite best treatment; f. treatment interruption for >=8 days during Cycle 0; Cycle 1 required by E7090-related toxicity, except for treatment interruption for >=8 days for reasons other than toxicity.
Time Frame: Cycle 0 (Cycle length= 7 days) up to Cycle 1 (Cycle length= 28 days)
Population: The DLT analysis set was the group of participants in the Part 1 who completed Cycle 0 and Cycle 1 treatment of E7090 with at least 75% compliance and were evaluated for DLT, and those who developed DLT during Cycle 0 or Cycle 1. This outcome measure was planned to be analyzed for Part 1 only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: E7090 1 mg With Solid Tumor | Part 1: E7090 2 mg With Solid Tumor | Part 1: E7090 4 mg With Solid Tumor | Part 1: E7090 8 mg With Solid Tumor | Part 1: E7090 16 mg With Solid Tumor | Part 1: E7090 30 mg With Solid Tumor | Part 1: E7090 60 mg With Solid Tumor | Part 1: E7090 100 mg With Solid Tumor | Part 1: E7090 140 mg With Solid Tumor | Part 1: E7090 180 mg With Solid Tumor
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: A TEAE was defined as an adverse event (AE) that emerged during the time from the first dose of study drug to 30 days following the last dose of study drug, having been absent at pretreatment (Baseline) or reemerged during treatment, having been present at pretreatment (Baseline) but stopped before treatment, or worsened in severity during treatment relative to the pretreatment state, when the AE was continuous. A Serious AE is any untoward medical occurrence that at any dose: resulted in death; was life threatening (that is, the participant was at immediate risk of death from the AE as it occurred; this does not include an event that, had it occurred in a more severe form or was allowed to continue, might have caused death) required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect or is medically important due to other reasons than the above mentioned criteria.
Time Frame: From the start of study drug administration up to 2 year 9 months
Population: The safety analysis set was the group of participants who received at least 1 dose of E7090. This outcome measure was planned to be analyzed for Part 1 and Part 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: E7090 1 mg With Solid Tumor | Part 1: E7090 2 mg With Solid Tumor | Part 1: E7090 4 mg With Solid Tumor | Part 1: E7090 8 mg With Solid Tumor | Part 1: E7090 16 mg With Solid Tumor | Part 1: E7090 30 mg With Solid Tumor | Part 1: E7090 60 mg With Solid Tumor | Part 1: E7090 100 mg With Solid Tumor | Part 1: E7090 140 mg With Solid Tumor | Part 1: E7090 180 mg With Solid Tumor | Part 2: E7090 140 mg With Gastric Cancer | Part 2: E7090 140 mg With Cholangiocarcinoma
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 3 | 10 | 6
Participants
  TEAEs | 2 | 1 | 1 | 2 | 2 | 2 | 3 | 3 | 3 | 3 | 10 | 6
  SAEs | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 1

3. Secondary Outcome: Part 2: Overall Survival (OS)
Description: OS was defined as the time from the date of first dose to the date of death from any cause. OS was estimated by using Kaplan-Meier method.
Time Frame: From the date of first dose of study drug up to 2 years and 8 months
Population: The efficacy analysis set was the group of participants who received at least 1 dose of E7090 and had both baseline and at least 1 post-baseline tumor assessments. This outcome measure was planned to be analyzed for Part 2 only.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2: E7090 140 mg With Gastric Cancer | Part 2: E7090 140 mg With Cholangiocarcinoma
Number analyzed (Participants) | 9 | 6
months | 4.27 [2.23 to 7.95] | 22.49 [6.37 to NA] — Upper limit of confidence interval could not be estimated due to an insufficient number of events.

4. Secondary Outcome: Part 2: Progression- Free Survival (PFS)
Description: PFS was defined as the time from the date of first dose to the first documented date of event (disease progression or death from any cause, whichever occurs first). PD was defined as at least a 20 percent (%) increase in the sum of LD of target and non-target lesions as compared with the smallest sum of long diameter (LD) and the increase of LD was at least 5 millimeter (mm) (including new lesions). The tumor assessment is based on Response Evaluation Criteria in Solid Tumor (RECIST) 1.1 criteria and was estimated using Kaplan-Meier method.
Time Frame: From the date of first dose of study drug up to 2 years and 8 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2: E7090 140 mg With Gastric Cancer | Part 2: E7090 140 mg With Cholangiocarcinoma
Number analyzed (Participants) | 9 | 6
months | 3.25 [0.95 to 4.86] | 8.26 [3.84 to NA] — Upper limit of confidence interval could not be estimated due to an insufficient number of events.

5. Secondary Outcome: Best Overall Response (BOR)
Description: Tumor assessment (target lesion, non-target lesion, and presence or absence of new lesion) was performed based on RECIST v1.1. Tumor marker was also measured. FDG-PET CT (fluorodeoxyglucose- Positron emission tomography computed tomography) also evaluated. Best overall responses were complete response (CR), partial response (PR), stable disease (SD), progression of disease (PD), and not evaluable (NE). CR was defined as disappearance of all target lesions and non-target lesions (a short diameter is <10 mm if it exists in a lymph node). PR was defined as at least 30% decrease in the sum of the LD of all target lesions, as compared with baseline summed LD. SD was defined as no known evidence of progressive disease or new bone lesions where SD was achieved at >=7 weeks after first dose.
Time Frame: From the date of first dose of study drug up to 2 years and 8 months
Population: The efficacy analysis set was the group of participants who received at least 1 dose of E7090 and had both baseline and at least 1 post-baseline tumor assessments. This outcome measure was planned to be analyzed for Part 1 and Part 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: E7090 1 mg With Solid Tumor | Part 1: E7090 2 mg With Solid Tumor | Part 1: E7090 4 mg With Solid Tumor | Part 1: E7090 8 mg With Solid Tumor | Part 1: E7090 16 mg With Solid Tumor | Part 1: E7090 30 mg With Solid Tumor | Part 1: E7090 60 mg With Solid Tumor | Part 1: E7090 100 mg With Solid Tumor | Part 1: E7090 140 mg With Solid Tumor | Part 1: E7090 180 mg With Solid Tumor | Part 2: E7090 140 mg With Gastric Cancer | Part 2: E7090 140 mg With Cholangiocarcinoma
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 3 | 9 | 6
Participants
  Complete Response (CR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response (PR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 5
  Stable Disease (SD) | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 4 | 1
  Progressive Disease (PD) | 1 | 2 | 1 | 2 | 1 | 1 | 2 | 2 | 1 | 1 | 4 | 0
  Not Evaluable (NE) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

6. Secondary Outcome: Part 2: Objective Response Rate (ORR)
Description: ORR was defined as a percentage of participants with BOR of CR or PR. ORR was assessed using RECIST 1.1. CR was defined as disappearance of all target lesions and non-target lesions (a short diameter is <10 mm if it exists in a lymph node). PR was defined as at least 30% decrease in the sum of the LD of all target lesions, as compared with baseline summed LD.
Time Frame: From screening up to 2 years and 8 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: E7090 140 mg With Gastric Cancer | Part 2: E7090 140 mg With Cholangiocarcinoma
Number analyzed (Participants) | 9 | 6
percentage of participants | 11.1 [0.3 to 48.2] | 83.3 [35.9 to 99.6]

7. Secondary Outcome: Part 2: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants with BOR of CR, PR or SD. DCR was assessed based on RECIST 1.1. CR was defined as disappearance of all target lesions and non-target lesions (a short diameter is <10 mm if it exists in a lymph node). PR was defined as at least 30% decrease in the sum of the LD of all target lesions, as compared with Baseline summed LD. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. SD was defined as no known evidence of progressive disease or new bone lesions where SD was achieved at >= 7 weeks after first dose.
Time Frame: From the date of first dose of study drug up to 2 years and 8 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: E7090 140 mg With Gastric Cancer | Part 2: E7090 140 mg With Cholangiocarcinoma
Number analyzed (Participants) | 9 | 6
percentage of participants | 55.6 [21.2 to 86.3] | 100.0 [54.1 to 100.0]

8. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for E7090
Time Frame: Part 1: Cycle 0 Day 1: 0-72 hours post dose (Cycle 0 is 7 days); Part 2: Cycle 1 Day 1: 0-24 hours post dose; (Cycle 1 is 28 days)
Population: The pharmacokinetic (PK) analysis set was the group of participants who received at least 1 dose of E7090 and had sufficient PK data to derive at least 1 PK parameter. This outcome measure was planned to be analyzed for Part 1 and Part 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part 1: E7090 1 mg With Solid Tumor | Part 1: E7090 2 mg With Solid Tumor | Part 1: E7090 4 mg With Solid Tumor | Part 1: E7090 8 mg With Solid Tumor | Part 1: E7090 16 mg With Solid Tumor | Part 1: E7090 30 mg With Solid Tumor | Part 1: E7090 60 mg With Solid Tumor | Part 1: E7090 100 mg With Solid Tumor | Part 1: E7090 140 mg With Solid Tumor | Part 1: E7090 180 mg With Solid Tumor | Part 2: E7090 140 mg With Gastric Cancer | Part 2: E7090 140 mg With Cholangiocarcinoma
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 2 | 10 | 6
nanogram per milliliter (ng/mL) | NA (NA) — The plasma concentrations of E7090 were below the limit of quantification at 1 mg dose in participants with solid tumors; therefore, Cmax could not be calculated. | NA (NA) — The plasma concentrations of E7090 were below the limit of quantification at 2 mg dose in participants with solid tumors; therefore, Cmax could not be calculated. | 1.27 (112) | 2.89 (4.41) | 8.54 (86.7) | 23.9 (98.1) | 38.5 (11.9) | 82.5 (34.9) | 206 (58.7) | 140 (34.6) | 188 (53.2) | 59.4 (107)

9. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for E7090
Time Frame: as for outcome 8
Population: The PK analysis set was the group of participants who received at least 1 dose of E7090 and had sufficient PK data to derive at least 1 PK parameter. This outcome measure was planned to be analyzed for Part 1 and Part 2.
Measure: Median (Full Range); unit: hour
Arm/Group | Part 1: E7090 1 mg With Solid Tumor | Part 1: E7090 2 mg With Solid Tumor | Part 1: E7090 4 mg With Solid Tumor | Part 1: E7090 8 mg With Solid Tumor | Part 1: E7090 16 mg With Solid Tumor | Part 1: E7090 30 mg With Solid Tumor | Part 1: E7090 60 mg With Solid Tumor | Part 1: E7090 100 mg With Solid Tumor | Part 1: E7090 140 mg With Solid Tumor | Part 1: E7090 180 mg With Solid Tumor | Part 2: E7090 140 mg With Gastric Cancer | Part 2: E7090 140 mg With Cholangiocarcinoma
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 2 | 10 | 6
hour | NA [NA to NA] — The plasma concentrations of E7090 were below the limit of quantification at 1 mg dose in participants with solid tumors; therefore, Tmax could not be calculated. | NA [NA to NA] — The plasma concentrations of E7090 were below the limit of quantification at 2 mg dose in participants with solid tumors; therefore, Tmax could not be calculated. | 1.51 [1.00 to 2.02] | 2.96 [2.92 to 3.00] | 2.01 [1.02 to 3.00] | 3.04 [0.93 to 5.15] | 3.00 [2.97 to 4.98] | 4.95 [2.97 to 5.10] | 4.88 [3.00 to 5.08] | 3.48 [1.95 to 5.00] | 2.96 [1.90 to 5.07] | 3.97 [2.95 to 4.98]

10. Secondary Outcome: AUC(0-24h): Area Under the Plasma Concentration-time Curve From Zero Time to 24 Hours
Time Frame: Part 1: Cycle 0 Day 1: 0-24 hours post dose (Cycle 0 is 7 days); Part 2: Cycle 1 Day 1: 0-24 hours post dose (Cycle 1 is 28 days)
Population: The PK analysis set was the group of participants who received at least 1 dose of E7090 and had sufficient PK data to derive at least 1 PK parameter. Here "overall number of participants analyzed" are those who were evaluable for this outcome measure. This outcome measure was planned to be analyzed for Part 1 and Part 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1: E7090 1 mg With Solid Tumor | Part 1: E7090 2 mg With Solid Tumor | Part 1: E7090 4 mg With Solid Tumor | Part 1: E7090 8 mg With Solid Tumor | Part 1: E7090 16 mg With Solid Tumor | Part 1: E7090 30 mg With Solid Tumor | Part 1: E7090 60 mg With Solid Tumor | Part 1: E7090 100 mg With Solid Tumor | Part 1: E7090 140 mg With Solid Tumor | Part 1: E7090 180 mg With Solid Tumor | Part 2: E7090 140 mg With Gastric Cancer | Part 2: E7090 140 mg With Cholangiocarcinoma
Number analyzed (Participants) | 2 | 2 | 1 | 1 | 2 | 2 | 3 | 3 | 3 | 2 | 10 | 6
h*ng/mL | NA (NA) — The plasma concentrations of E7090 were below the limit of quantification at 1 mg dose in participants with solid tumors; therefore, AUC(0-24h) could not be calculated. | NA (NA) — The plasma concentrations of E7090 were below the limit of quantification at 2 mg dose in participants with solid tumors; therefore, AUC(0-24h) could not be calculated. | 5.71 (NA) — As only one participant was present, Standard Deviation could not be calculated. | 19.8 (NA) — As only one participant was present, Standard Deviation could not be calculated. | 55.1 (45.2) | 164 (39.4) | 341 (31.2) | 788 (52.2) | 2100 (80.5) | 1760 (50.4) | 1590 (70.5) | 618 (87.7)

11. Secondary Outcome: Part 1: CL/F: Apparent Total Clearance for E7090
Time Frame: Part 1: Cycle 0 Day 1: 0-72 hours post dose (Cycle 0 is 7 days)
Population: The PK analysis set was the group of participants who received at least 1 dose of E7090 and had sufficient PK data to derive at least 1 PK parameter. This outcome measure was planned to be analyzed for Part 1 only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/h)
Arm/Group | Part 1: E7090 1 mg With Solid Tumor | Part 1: E7090 2 mg With Solid Tumor | Part 1: E7090 4 mg With Solid Tumor | Part 1: E7090 8 mg With Solid Tumor | Part 1: E7090 16 mg With Solid Tumor | Part 1: E7090 30 mg With Solid Tumor | Part 1: E7090 60 mg With Solid Tumor | Part 1: E7090 100 mg With Solid Tumor | Part 1: E7090 140 mg With Solid Tumor | Part 1: E7090 180 mg With Solid Tumor
Number analyzed (Participants) | 2 | 2 | 1 | 2 | 2 | 2 | 3 | 3 | 3 | 2
Liter per hour (L/h) | NA (NA) — The plasma concentrations of E7090 were below the limit of quantification at 1 mg dose in participants with solid tumors; therefore, CL/F could not be calculated. | NA (NA) — The plasma concentrations of E7090 were below the limit of quantification at 2 mg dose in participants with solid tumors; therefore, CL/F could not be calculated. | 700 (NA) — As only one participant was present, Standard Deviation could not be calculated. | NA (NA) — CL/F could not be calculated as at least 3 concentration points in the terminal phase were not available due to being below the limit of quantification. | 243 (60.2) | 126 (14.6) | 116 (41.2) | 95.5 (48.8) | 46.7 (109) | 66.7 (41.8)

ADVERSE EVENTS:
Time Frame: From the start of study drug administration up to 2 year and 9 months
Arm/Group | Part 1: E7090 1 mg With Solid Tumor | Part 1: E7090 2 mg With Solid Tumor | Part 1: E7090 4 mg With Solid Tumor | Part 1: E7090 8 mg With Solid Tumor | Part 1: E7090 16 mg With Solid Tumor | Part 1: E7090 30 mg With Solid Tumor | Part 1: E7090 60 mg With Solid Tumor | Part 1: E7090 100 mg With Solid Tumor | Part 1: E7090 140 mg With Solid Tumor | Part 1: E7090 180 mg With Solid Tumor | Part 2: E7090 140 mg With Gastric Cancer | Part 2: E7090 140 mg With Cholangiocarcinoma
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/3 | 0/3 | 0/3 | 0/3 | 10/10 | 5/6
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 2/2 | 0/2 | 1/2 | 0/3 | 0/3 | 0/3 | 0/3 | 4/10 | 1/6
Other Adverse Events (participants affected / at risk) | 2/2 | 1/2 | 1/2 | 2/2 | 2/2 | 2/2 | 3/3 | 3/3 | 3/3 | 3/3 | 10/10 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: E7090 1 mg With Solid Tumor (N=2) | Part 1: E7090 2 mg With Solid Tumor (N=2) | Part 1: E7090 4 mg With Solid Tumor (N=2) | Part 1: E7090 8 mg With Solid Tumor (N=2) | Part 1: E7090 16 mg With Solid Tumor (N=2) | Part 1: E7090 30 mg With Solid Tumor (N=2) | Part 1: E7090 60 mg With Solid Tumor (N=3) | Part 1: E7090 100 mg With Solid Tumor (N=3) | Part 1: E7090 140 mg With Solid Tumor (N=3) | Part 1: E7090 180 mg With Solid Tumor (N=3) | Part 2: E7090 140 mg With Gastric Cancer (N=10) | Part 2: E7090 140 mg With Cholangiocarcinoma (N=6)
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour obstruction (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombophlebitis migrans (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: E7090 1 mg With Solid Tumor (N=2) | Part 1: E7090 2 mg With Solid Tumor (N=2) | Part 1: E7090 4 mg With Solid Tumor (N=2) | Part 1: E7090 8 mg With Solid Tumor (N=2) | Part 1: E7090 16 mg With Solid Tumor (N=2) | Part 1: E7090 30 mg With Solid Tumor (N=2) | Part 1: E7090 60 mg With Solid Tumor (N=3) | Part 1: E7090 100 mg With Solid Tumor (N=3) | Part 1: E7090 140 mg With Solid Tumor (N=3) | Part 1: E7090 180 mg With Solid Tumor (N=3) | Part 2: E7090 140 mg With Gastric Cancer (N=10) | Part 2: E7090 140 mg With Cholangiocarcinoma (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 4 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Serous retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Macular oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Corneal disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subretinal fluid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 2 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 3 | 2 | 4
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1
Angular cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Glossitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 2
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mucosal haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 3 | 1 | 3 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 3 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fibrin D dimer increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 10 | 6
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 4 | 2
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Paralysis recurrent laryngeal nerve (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 4 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 4
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/10/NCT02275910/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-26): https://cdn.clinicaltrials.gov/large-docs/10/NCT02275910/SAP_001.pdf